CLINICAL TRIAL: NCT04516395
Title: Optimizing Antibiotic Dosing Regimens for the Treatment of Infection Caused by Carbapenem Resistant Enterobacteriaceae: the Study of in Vitro Activity of Monotherapy and Combination Therapy, PK/PD Study and Treatment Outcomes
Brief Title: Optimizing Antibiotic Dosing Regimens for the Treatment of Infection Caused by Carbapenem Resistant Enterobacteriaceae
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Q011h/63
Record Dates: First submitted 2020-07-20; First posted 2020-08-18 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Drug Resistance; Carbapenem-Resistant Enterobacteriaceae Infection; Sepsis; Septic Shock; Critical Illness; Clinical Outcomes; Treatment Outcomes
Keywords: Pharmacokinetics/Pharmacodynamics; Antibiotic combination regimens; Dose-optimization; Carbapenem-Resistant Enterobacteriaceae Infection
MeSH Terms: conditions — Sepsis; Shock, Septic; Critical Illness

STUDY DESIGN:
Intervention Model Description: According to the model, it divided into two parts - retrospective chart review and prospective data collection. Single independent patient group will be divided two parts depending on over a period of time. The patients in the retrospective part received a standard treatment become a control group, while the patients in the prospective part received the intervention become an experimental group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimal antibiotic combination regimens (Experimental): The patients in the groups will be given the optimal antibiotic combination regimens.
  Interventions: Other: Combined antibiotic regimens
- Standard antibiotic regimens (Other): The patients in the groups will be given the standard antibiotic regimens.
  Interventions: Other: Standard antibiotic regimens

INTERVENTIONS:
Other: Combined antibiotic regimens — Combined antibiotic combinations defined as the optimal antibiotic combination regimens which are created from in vitro study and the application of PK/PD.
  Arms: Optimal antibiotic combination regimens
Other: Standard antibiotic regimens — Standard antibiotic regimens defined as the antibiotic regimens which are generally given to the patients following to the hospital protocol.
  Arms: Standard antibiotic regimens

SUMMARY:
The purpose of this study is to evaluate the treatment outcomes in patients with CRE infections.

DETAILED DESCRIPTION:
Antibiotic resistance is one of the major problems because of global burden. Resistant pathogens are non-susceptible to available antibiotics, causing of high clinical mortality (clinical impact) and high budget (economic impact), whereas new antibiotics in drug development are fewer. Carbapenem-Resistant Enterobacteriaceae (CRE) are categorized into one of the critical groups in World Health Organization's lists. In Thailand, the spread of CRE have been risen continuously since 2011.

Diverse actions are designed to address antibiotic resistance with limited resources, known as antimicrobial stewardship programs (ASPs). Dose-optimization by using PK/PD (Pharmacokinetics/Pharmacodynamics) application is recommendation of supplemental strategies in clinical routine practice. The benefit of the strategy is to reduce inappropriate antibiotic use and provide minimum resistance as well as maximum the success of clinical treatment.

Antibiotic combination regimens have a role for the CRE treatment. However, current evidence in clinical study is not concluded which the best or optimal combined antibiotics are. The reasons may be that combined antibiotics often vary among different sites of infection, causative pathogens, the patterns of local antimicrobial susceptibility and patient comorbidity. As the results, the antibiotic combination regimens for the treatment any infections caused by CRE is needed for further investigation. The anticipated result is to fill the limited data of the appropriate antibiotic regimens for individual Thai patients.

ELIGIBILITY:
Inclusion Criteria:

1. Any patients are diagnosed any diseases caused by CRE infection by physicians at Phramongkutklao hospital during 1/4/2018 to 30/4/2021.
2. Any patients are more than 18 years old.
3. Any patients have at least 1 criterion as following 3.1 Any patients have at least 2 of the signs and symptoms of Systemic inflammatory response syndrome (SIRS), including

   * Fever (temperature > 38 °C) or hypothermia (temperature < 36°C)
   * Tachypnea (heart rate > 90 beats per minute)
   * Respiratory rate > 20 beats per minute or Paco2 < 32 mm Hg (4.3 kPa)
   * White blood cell count > 12,000 cells per millilitre (leukocytosis) or < 4,000 cells per milliliter (leukopenia) 3.2. Any patients are diagnosed with sepsis or have ≥ 2 points of Sequential Organ Failure Assessment (SOFA) Score or qSOFA (Quick SOFA) Score.

3.3. Any patients are diagnosed with septic shock or are received vasopressors (eg, dopamine, norepinephrine, epinephrine, vasopressin, phenylephrine), mean arterial pressure (MAP) < 65 mm Hg, and lactate > 2 mmol/L (18 mg/dL) 3.4 Any patients are received mechanical ventilation 3.5 Any patients are admitted at ICU ward.

Exclusion Criteria:

1. Patients are breast-feeding or pregnancy.
2. Patients are insufficient or incomplete information on the medical electronic record such as patients transferred.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement or failure | up to 8 weeks
  * Clinical improvement was defined as resolution of the signs and symptoms of the infection with no change or addition antibiotic therapy at the end of treatment course, excepting de-escalation to a narrower spectrum antibiotic.
  * Clinical failure was defined as the signs and symptoms of the infection being more serious with change or addition antibiotic therapy against CRE.

SECONDARY OUTCOMES:
Mortality | Within 14 and 28/30 days after discharge
  All cause mortality
Length of stay | up to 12 weeks
  The duration of a hospitalization
Physician acceptance rates | up to 72 hours after reporting the bacterial culture results
  The rates of physicians' acceptance of an recommended optimal regimen
Microbiological outcomes | Before discharge
  Bacterial response in cultures after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wichai Santimaleeworagun, Principal Investigator — Silpakorn University
Locations (1):
- Phramongkutklao hospital, Bangkok, Thailand

REFERENCES:
- [Result] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Result] Tillotson G. A crucial list of pathogens. Lancet Infect Dis. 2018 Mar;18(3):234-236. doi: 10.1016/S1473-3099(17)30754-5. Epub 2017 Dec 21. No abstract available. PMID 29276050
- [Result] Barlam TF, Cosgrove SE, Abbo LM, MacDougall C, Schuetz AN, Septimus EJ, Srinivasan A, Dellit TH, Falck-Ytter YT, Fishman NO, Hamilton CW, Jenkins TC, Lipsett PA, Malani PN, May LS, Moran GJ, Neuhauser MM, Newland JG, Ohl CA, Samore MH, Seo SK, Trivedi KK. Implementing an Antibiotic Stewardship Program: Guidelines by the Infectious Diseases Society of America and the Society for Healthcare Epidemiology of America. Clin Infect Dis. 2016 May 15;62(10):e51-77. doi: 10.1093/cid/ciw118. Epub 2016 Apr 13. PMID 27080992
- [Result] Asin-Prieto E, Rodriguez-Gascon A, Isla A. Applications of the pharmacokinetic/pharmacodynamic (PK/PD) analysis of antimicrobial agents. J Infect Chemother. 2015 May;21(5):319-29. doi: 10.1016/j.jiac.2015.02.001. Epub 2015 Feb 12. PMID 25737147
- [Result] Rodriguez-Bano J, Gutierrez-Gutierrez B, Machuca I, Pascual A. Treatment of Infections Caused by Extended-Spectrum-Beta-Lactamase-, AmpC-, and Carbapenemase-Producing Enterobacteriaceae. Clin Microbiol Rev. 2018 Feb 14;31(2):e00079-17. doi: 10.1128/CMR.00079-17. Print 2018 Apr. PMID 29444952
- [Result] Tamma PD, Goodman KE, Harris AD, Tekle T, Roberts A, Taiwo A, Simner PJ. Comparing the Outcomes of Patients With Carbapenemase-Producing and Non-Carbapenemase-Producing Carbapenem-Resistant Enterobacteriaceae Bacteremia. Clin Infect Dis. 2017 Feb 1;64(3):257-264. doi: 10.1093/cid/ciw741. Epub 2016 Nov 9. PMID 28013264
- [Result] Demidenko E, Miller TW. Statistical determination of synergy based on Bliss definition of drugs independence. PLoS One. 2019 Nov 25;14(11):e0224137. doi: 10.1371/journal.pone.0224137. eCollection 2019. PMID 31765385
- [Result] Sheu CC, Chang YT, Lin SY, Chen YH, Hsueh PR. Infections Caused by Carbapenem-Resistant Enterobacteriaceae: An Update on Therapeutic Options. Front Microbiol. 2019 Jan 30;10:80. doi: 10.3389/fmicb.2019.00080. eCollection 2019. PMID 30761114
- [Result] Gutierrez-Gutierrez B, Salamanca E, de Cueto M, Hsueh PR, Viale P, Pano-Pardo JR, Venditti M, Tumbarello M, Daikos G, Canton R, Doi Y, Tuon FF, Karaiskos I, Perez-Nadales E, Schwaber MJ, Azap OK, Souli M, Roilides E, Pournaras S, Akova M, Perez F, Bermejo J, Oliver A, Almela M, Lowman W, Almirante B, Bonomo RA, Carmeli Y, Paterson DL, Pascual A, Rodriguez-Bano J; REIPI/ESGBIS/INCREMENT Investigators. Effect of appropriate combination therapy on mortality of patients with bloodstream infections due to carbapenemase-producing Enterobacteriaceae (INCREMENT): a retrospective cohort study. Lancet Infect Dis. 2017 Jul;17(7):726-734. doi: 10.1016/S1473-3099(17)30228-1. Epub 2017 Apr 22. PMID 28442293